CLINICAL TRIAL: NCT01650103
Title: Hemodynamic Indexes and Renal Perfusion: Indirect Evaluation of Blood Volume Using the Association Between ScvO2 and Urinary Electrolytes in Patients Undergoing Major Surgery.
Brief Title: Evaluation of Hemodynamics and Amount of Blood Flowing Through the Kidneys by Measuring Some Physiological Substances in Blood and Urines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Dr. Paolo Feltracco, Principal Investigator, Azienda Ospedaliera di Padova
Other Study IDs: 2660P
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Hypovolemia; Renal Hypoperfusion
Keywords: hypovolemia; renal hypoperfusion; major surgery; sodium; potassium; chloride; ScvO2; hemodynamic indexes
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to verify any existing relationship between mixed oxygen saturation (from central venous catheter) and urinary sodium, potassium, chloride in determining the volemic state and renal perfusion of patients undergoing major surgical interventions.

ELIGIBILITY:
Inclusion Criteria:

* thoracic-abdominal major surgical operations
* placing of a central venous catheter and urinary catheter
* age 18-75
* ASA class I-III

Exclusion Criteria:

* age above 75 or under 18
* ASA class IV
* trauma, sepsis and/or heart-lung failure
* liver transplantation
* kidney transplantation
* pre-existing renal failure
* pregnant patients
* patients unable to give their written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Determination of mixed oxygen saturation in central venous blood (ScvO2) and three urinary electrolytes (sodium, potassium, chloride) | During the stay of the patient in the operating room (in average 6 hours) and the eventual stay in the post-surgery intensive care unit (in average 1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ori, Prof. M.D., Study Chair — University of Padova; Paolo Feltracco, M.D., Principal Investigator — Azienda Ospedaliera di Padova; Andrea Bortolato, M.D., Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Padova, Italy